CLINICAL TRIAL: NCT05103241
Title: Single-center, Open-label, Non-randomized and Single-dose Clinical Trial to Explore the Mass Balance of Oral Suspension of 40 mg/100 μCi [14C]GP681 in Healthy Chinese Male Volunteers
Brief Title: A Phase I Mass Balance Study of [14C]GP681 in Healthy Chinese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRC-C2131
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Open-label, radiolabeled, single-dose study of an oral solution of [14C]GP681(40mg/100μCi) in 6 healthy male volunteer.
Masking Description: Nonrandomized and open labeled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]GP681 (Experimental): Subject will receive single dose of orally [14C] GP681 .
  Interventions: Drug: [14C] GP681

INTERVENTIONS:
Drug: [14C] GP681 — 40 mg suspension containing 100μCi of [14C]GP681

SUMMARY:
This study is a single-center, open-label, and single-dose clinical study to evaluate the mass balance, biotransformation and pharmacokinetics of [14C]GP681 in healthy Chinese male volunteers, revealing the overall pharmacokinetic characteristics of GP681 in humans, and providing a reference for the rational administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 40years, inclusive;
2. A history of regular bowel movements (average 1or 2 bowel movements per day)
3. Body weight ≥50.0 kg and body mass index (BMI) between19-26 kg/m^2(inclusive);
4. Normal physical examination, vital signs, 12-lead ECG, Chest X-ray images (anteroposterior) and clinical laboratory values, or any abnormality that is non-clinically significant;
5. Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for at least half a year after the final dose of study drug
6. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions.

Exclusion Criteria:

1. History of allergic conditions or allergic diseases, or a history of allergic reactions attributed to GP681 or any of the ingredients of its formulation or similar drugs. Those who cannot follow a uniform diet for special dietary requirements.
2. Subjects with swallowing difficulties, or have diseases such as hemorrhoids, perianal diseases with regular/bleeding in the stool, habitual constipation or diarrhea, irritable bowel syndrome and inflammatory bowel diseases, affecting drug absorption, distribution, metabolism, excretion or the efficacy and safety of the drug.
3. History of gastrointestinal ulcer or bleeding; Or history of any clinically significant diseases or diseases which may affect the result of this study, such as gastrointestinal, circulatory, respiratory, endocrine, neurological, urinary, hematological, immunological, psychiatric and metabolic diseases;
4. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade de pointes ventricular tachycardia, ventricular tachycardia, prolonged QT syndrome, or symptoms of prolonged QT syndrome and family history;
5. Patients who have undergone surgery within 6 months before the screening period, or who have undergone major surgery within 28 days, or whose surgical incision is not completely healed; Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury;
6. Any positive test result of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
7. Received any drugs that inhibit or induce the CYP450 enzyme (i.e., inducers-barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors- SSRI-antidepressant, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines) 30 days prior to screening period;
8. Received any drugs (including Chinese herbal medicine, vitamins and supplements) within 14 days prior to dosing, or participation in another clinical trial within 3 months before dosing.
9. Those who have lost blood or donated up to 400 mL within 3 months before dosing, or those who plan to donate blood within 1 month after the end of this study;
10. Smoking more than 10 cigarettes per day;
11. Average weekly intake of alcohol is more than 14 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) within the 6 months prior to dosing, or a positive ethanol breath test at screening;
12. Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.) in the 1 year prior to the screening period; Or screening for positive urine drug abuse (drug) tests;
13. Habitual or excessive consumption (more than 8 cups, 1cup=250mL) of grapefruit juice, tea, coffee and/or caffeinated beverages;
14. Workers engaged in conditions requiring long-term exposure to radioactivity; Or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before this study or have participated in the radiopharmaceutical labeling test;
15. Subjects with poor compliance, or not suitable for this study as judged by the investigator.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — age of 18-40 (inclusive)
Enrollment: 6 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
The distribution of GP681 in the whole blood and plasma, and the radioactive pharmacokinetics following the single orally administered [14C]GP681 in healthy Chinese male volunteers. | Up to 336 hours (approx) from the start of administration.
  The percentage of radioactive dose of [14C] radiolabelled GP681 recovered in blood and in total.
Quantitive analysis of whole radioactivity of excrement of orally administered [14C]GP681 in healthy Chinese male subjects to obtain the mass balance data and the main excretion pathway in human body. | Up to 432 hours (approx) from the start of administration.
  The percentage of radioactive dose of [14C] radiolabelled GP681 recovered in urine, faeces and in total.
Quantitive analysis of the concentrations of GP681 and its major metabolites (such as GP1707D07) in plasma using the validated LC-MS/MS to obtain pharmacokinetic data. | Up to 336 hours (approx) from the start of administration.
  The concentrations of GP681 and its major metabolites in plasma.
Identification of the main metabolites and biotransformation pathway of GP681 following the single orally administered [14C]GP681 in healthy Chinese male volunteers | Up to 432 hours (approx) from the start of administration.
  Proportion of different metabolites.
Evaluation of safety following the single orally administered [14C]GP681 in healthy Chinese male volunteers. | Up to 432 hours (approx) from the start of administration.
  Adverse events assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China